CLINICAL TRIAL: NCT04674306
Title: Phase I Trial of Adjuvant Therapy With an Alpha-lactalbumin Vaccine in Patients With Non-Metastatic Triple-Negative Breast Cancer at High Risk of Recurrence
Brief Title: Adjuvant Therapy With an Alpha-lactalbumin Vaccine in Triple-Negative Breast Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: George T. Budd (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Anixa Biosciences, Inc. (Unknown)
Responsible Party: Sponsor-Investigator, George T. Budd, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE6119; W81XWH-17-1-0593 (Other Grant/Funding Number: United States Department of Defense); W81XWH-17-1-0592 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2020-12-13; First posted 2020-12-19 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Pathologic Stage IIA-IIIC Triple-Negative Breast Cancer; TNBC - Triple-Negative Breast Cancer; Residual Disease
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Neoplasm, Residual | interventions — Zymosan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment α-lactalbumin and zymosan (Experimental): Participants diagnosed with triple negative breast cancer will be treated with successively higher doses of α-lactalbumin and zymosan in a 3 + 3 trial design. Treatment will involve 3 vaccinations every 2 weeks. Participants will be enrolled into 1 of 5 different dose levels each comprised of cohorts of 1-6 participants until the MTD has been identified (intra-patient dose escalation not permitted), after which the MTD will be expanded to 6 participants. Successively lower doses will be expanded to 6 participants until the lowest DL associated with immune response has been expanded.
  DL1: 10 mcg a-lactalbumin + 10 mcg Zymosan Original DL2:100 mcg a-lactalbumin + 100 mcg Zyomsan DL2: 100 mcg a-lactalbumin + 10 mcg Zyomsan DL3: 500 mcg a-lactalbumin + 10 mcg Zymosan DL1b: 50 mcg a-lactalbumin + 10 mcg Zymosan DL1e: 10 mcg a-lactalbumin + 20 mcg Zymosan DL1f: 20 mcg a-lactalbumin + 10 mcg Zymosan DL1g: 20 mcg a-lactalbumin + 10 mcg Zymosan (if DL1e is too toxic)
  Interventions: Biological: α-lactalbumin vaccine; Biological: Zymosan
- Preventitive a-lactalbumin and zymosan (Experimental): Participants with a genetic risk for developing TNBC who plan to undergo prophylactic mastectomy will be treated with α-lactalbumin and zymosan at doses based on the TNBC cohort. Treatment will involve 3 vaccinations every 2 weeks. Participants enrolled in the prevention cohort will be enrolled at the dose level being used in the TNBC cohort if no DLTs above Grade 1 have been observed. If the TNBC cohort proceeds to the next dose level before another prevention cohort patient is enrolled, the next prevention patient will be enrolled on the next dose level along with the TNBC cohort.
  DL1: 10 mcg a-lactalbumin + 10 mcg Zymosan Original DL2:100 mcg a-lactalbumin + 100 mcg Zyomsan DL2: 100 mcg a-lactalbumin + 10 mcg Zyomsan DL3: 500 mcg a-lactalbumin + 10 mcg Zymosan DL1b: 50 mcg a-lactalbumin + 10 mcg Zymosan DL1e: 10 mcg a-lactalbumin + 20 mcg Zymosan DL1f: 20 mcg a-lactalbumin + 10 mcg Zymosan DL1g: 20 mcg a-lactalbumin + 10 mcg Zymosan (if DL1e is too toxic)
  Interventions: Biological: α-lactalbumin vaccine; Biological: Zymosan
- Standard of Care with a-lactalbumin and zymosan (Experimental): Participants undergoing chemo-immunotherapy for operable triple-negative breast cancer will be treated with α-lactalbumin concurrently with standard of care adjuvant pembrolizumab after having completed all pre- and postoperative chemotherapy and radiation therapy, with the exception of Xeloda/capecitabine at provider discretion. Treatment will involve 3 vaccinations every 2 weeks. Participants enrolled in the Pembrolizumab cohort will be enrolled at the proper Optimal Immunologic Dose as defined by the TNBC and preventative cohorts and based on information available at the time of study entry.
  DL1: 10 mcg a-lactalbumin + 10 mcg Zymosan Original DL2:100 mcg a-lactalbumin + 100 mcg Zyomsan DL2: 100 mcg a-lactalbumin + 10 mcg Zyomsan DL3: 500 mcg a-lactalbumin + 10 mcg Zymosan DL1b: 50 mcg a-lactalbumin + 10 mcg Zymosan DL1e: 10 mcg a-lactalbumin + 20 mcg Zymosan DL1f: 20 mcg a-lactalbumin + 10 mcg Zymosan DL1g: 20 mcg a-lactalbumin + 10 mcg Zymosan (if DL1e is too toxic)
  Interventions: Biological: α-lactalbumin vaccine; Biological: Zymosan

INTERVENTIONS:
Biological: α-lactalbumin vaccine — α-lactalbumin vaccine will be administered subcutaneously in rotating sites (vaccine will not be administered in the arms of any participant, due to likelihood of prior bilateral mastectomy).
  DL1: 10 mcg
  DL Original 2: 100 mcg
  DL2: 100 mcg
  DL3: 500 mcg
  D1b: 50 mcg
  D1e: 10 mcg
  D1f: 20 mcg
  D1g: 20 mcg (D1g will only be utilized if D1c is deemed too toxic)
  Other Names: α-lactalbumin protein
Biological: Zymosan — Adjuvant used in vaccine preparation
  DL1: 10 mcg
  DL Original 2: 100 mcg
  DL2: 10 mcg
  DL3: 10 mcg
  D1b: 10 mcg
  D1e: 20 mcg
  D1f: 20 mcg
  D1g: 1o mcg (D1g will only be utilized if D1c is deemed too toxic)

SUMMARY:
The purpose of this study is to determine the safety as well as the most effective dose of the alpha-lactalbumin vaccine (aLA breast cancer vaccine) to treat patients with non-metastatic triple negative breast cancer, participants who are of cancer-free but may be at risk for triple-negative breast cancer, and for participants who are receiving adjuvant pembrolizumab following initial triple negative breast cancer treatment.

DETAILED DESCRIPTION:
This is an open-label, phase I dose-escalation trial that will be performed on three successive cohorts. The first cohort is comprised of participants with high-risk triple-negative breast cancer. The second is made up of participants scheduled to undergo bilateral prophylactic mastectomy due to their genetic risk of triple-negative breast cancer. The third cohort is comprised of participants who have had treatment for their triple-negative breast cancer treatment, receiving adjuvant pembrolizumab. These cohorts will be treated with successively higher doses of α-lactalbumin and zymosan.

This aLA breast cancer vaccine is an investigational (experimental) drug that the study team believes will work by stimulating the immune system to fight the participant's cancer, in a way similar to the way the immune system fights off an infection after a vaccination for that infection. α-lactalbumin Vaccine is experimental because it is not approved by the Food and Drug Administration (FDA).

A traditional "3+3" Phase I trial design will be employed for the cohorts to determined the Maximum Tolerated Dose (MTD). After identification of the MTD, if at least 1 participant has an immunologic response (correlative measurement), successively lower dose levels will be expanded to a total of 6 participants and immunologic response assessed. Enrollment will stop if a dose level is reached for which no responses are observed. Dose-Limiting toxicities (DLTs) in 2 or more of 6 participants, the next lower dose will be considered the new MTD.

Objectives are to determine MTD, DLT incidence, and Lowest Immunologic Dose (LID) for each cohort.

Toxicity will be assessed every 2 weeks until day 56 and at day 84 or at off-study. Participants will be offered participation in long-term follow-up involving contact or in-person follow-up for late toxicity and survival every 3 months for 2 years, every 6 months for an additional 3 years, and then annually for 10 years.

ELIGIBILITY:
Inclusion Criteria:

Triple Negative Cohort:

* Histologically proven invasive breast cancer.
* Primary tumor must be ER-negative (ER in <1% of cells), PR-negative (PR in <1% of cells), and HER2-negative (0-1+ by IHC or FISH ratio<2.0 with signal number <6/cell), or consistent with contemporary NCCN guidelines (https://www.nccn.org/).
* Patients must be high risk, defined as either:
* Pathologic stage IIA, IIB, IIIA, IIIB, or IIIC by AJCC 8, or
* Residual invasive cancer in breast or regional nodes following preoperative chemotherapy.
* Patients must have no convincing evidence of recurrent disease based on one of the following:
* bone scan and imaging scans of the chest/abdomen/pelvis or
* FDG PET scan.
* ≥1 months since last active therapy (chemotherapy, radiation therapy, or surgery) and ≤ 36 months since the initiation of treatment for the current cancer, based on the period of highest risk for patients with Stages I-III triplenegative breast cancer [33, 34].
* Treatment prior to enrollment must be consistent with NCCN guidelines extant at the time treatment was given, found at: https://www.nccn.org/.
* Age greater than or equal to 18 years.
* ECOG Performance Status 0-1.
* Adequate major organ function, defined as:

WBC ≥ 3,000/mcl, hemoglobin ≥ 10.0 gm/dL, platelets ≥ 100,000/mcL, total bilirubin within normal limits, ALT/AST <3 x upper limits of normal (ULN), serum creatinine ≤ 1.5 x ULN.

* Serum prolactin level must be ≤ upper limits of normal (ULN).
* Subjects must have the ability to understand and the willingness to sign and provide a written informed consent document.
* Subjects must have archival tissue available for potential correlative studies (e.g., assays for α-lactalbumin expression or tumor infiltrating lymphocytes), but tumors will not be required to exhibit overexpression of α-lactalbumin for enrollment.
* Subject agrees not to use alternative therapies from the time of informed consent through 30 days following the last vaccine injection. ). Patients may be asked to complete a "wash out" period prior to the first dose of vaccine at the PI's discretion to ensure the absence of all alternative therapies.

Prevention Cohort:

* Participant must have a high risk for developing triple-negative breast cancer, defined as: carrying a deleterious mutation in BRCA1, PALB2 or BRCA2
* Patients must have no evidence of breast cancer based on both of the following: Negative mammography or breast MRI within 180 days, Negative breast examination by a physician or advanced practice practitioner within 30 days
* Age ≥ 18 years
* ECOG Performance Status 0-1.
* Adequate major organ function, defined as: WBC ≥ 3,000/mcl, hemoglobin ≥ 10.0 gm/dL, platelets >100,000/mcL, total bilirubin within normal limits, ALT/AST <3 x upper limits of normal (ULN), serum creatinine ≤ 1.5 x ULN.
* Serum prolactin level must be ≤ upper limits of normal (ULN)
* Subjects must have the ability to understand and the willingness to sign and provide a written informed consent document.
* Subject agrees not to use alternative therapies from the time of informed consent through 30 days following the last vaccine injection. Patients may be asked to complete a "wash out" period prior to the first dose of vaccine at the PI's discretion to ensure the absence of all alternative therapies.

Pembrolizumab Cohort:

* Histologically proven invasive breast cancer.
* Primary tumor must be ER-negative (ER in <1% of cells), PR-negative (PR in <1% of cells), and HER2-negative (0-1+ by IHC or FISH ratio <2.0 with signal number <6/cell), or consistent with contemporary NCCN guidelines (https://www.nccn.org/).
* Patients must be high risk, defined as having residual invasive cancer in breast or regional nodes following pre-operative chemotherapy.
* Patients must have no convincing evidence of recurrent disease based on one of the following: Bone scan and imaging scans of the chest/abdomen/pelvis, or: FDG PET scan.
* >1 months since last active therapy with chemotherapy (excluding Xeloda/capecitabine), radiation therapy, or surgery and at least 6 weeks of pembrolizumab therapy planned after the first dose of alpha-lactalbumin vaccine.
* Treatment prior to enrollment must be consistent with NCCN guidelines extant at the time treatment was given, found at: https://www.nccn.org/.
* Age >18 years.
* ECOG Performance Status 0-1.
* Adequate major organ function, defined as: WBC > 3,000/mcl, hemoglobin > 10.0 gm/dL, platelets > 100,000/mcL, total bilirubin within normal limits, ALT/AST <3 x upper limits of normal (ULN), serum creatinine < 1.5 x ULN.
* Serum prolactin level must be < upper limits of normal (ULN).
* Subjects must have the ability to understand and the willingness to sign and provide a written informed consent document.
* Subjects must have archival tissue available for potential correlative studies (e.g., assays for α-lactalbumin expression or tumor infiltrating lymphocytes), but tumors will not be required to exhibit overexpression of α-lactalbumin for enrollment.
* Subject agrees not to use alternative therapies from the time of informed consent through 30 days following the last vaccine injection. Patients may be asked to complete a "wash out" period prior to the first dose of vaccine at the PI's discretion to ensure the absence of all alternative therapies.

Exclusion Criteria:

Triple Negative Cohort:

* Receipt of cytotoxic chemotherapy within 4 weeks of study entry (except for capecitabine in subjects enrolled in the pembrolizumab cohort).
* Radiation therapy within 4 weeks of study entry.
* Failure to recover from the toxicity of the previous therapy to CTCAE Grade 0-1, except for alopecia and grade 2 neuropathy.
* Need for systemic corticosteroid use (except as physiologic replacement, defined as prednisone 10 mg/day or equivalent).
* Need for immunosuppression (e.g., for a history of organ transplantation).
* Known HIV infection.
* Active or planned lactation or pregnancy.
* Patients taking or planning to take oral contraceptives will be excluded, as there is some evidence that such agents can induce lactational foci. This includes patients using hormone containing IUD's.
* Refusal to use effective non-hormonal contraception. Acceptable contraception methods include but may not be limited to barrier contraception (diaphragm or condom), non-hormonal intrauterine device, vasectomy of male partner.
* Subjects receiving any other investigational agents within the last 4 weeks.
* Subjects with any known recurrence or metastasis.
* Subjects with a history of another active invasive malignancy within 5 years of study entry.
* History of allergic reactions to α-lactalbumin, human milk (excluding lactose intolerance), zymosan, or other agents used in this study.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects with known hyperprolactinemia.
* Subjects being treated with drugs known to cause hyperprolactinemia
* Subjects diagnosed with TNBC while pregnant.
* Subjects having lactated within 6 months of study start (first dose of vaccine).

Prevention Cohort:

* Receipt of cytotoxic chemotherapy within 4 weeks of study entry (including for benign indications).
* Radiation therapy within 4 weeks of study entry (including for benign indications)
* Need for systemic corticosteroid use (except as physiologic replacement, defined as prednisone 10 mg/day or equivalent).
* Need for immunosuppression (e.g., for a history of organ transplantation).
* Known HIV infection.
* Active or planned lactation or pregnancy.
* Patients taking or planning to take oral contraceptives will be excluded, as there is some evidence that such agents can induce lactational foci. This includes patients using hormone containing IUD's.
* Refusal to use effective non-hormonal contraception. Acceptable contraception methods include but may not be limited to barrier contraception (diaphragm or condom), non-hormonal intrauterine device, vasectomy of male partner.
* Subjects receiving any other investigational agents within the last 4 weeks.
* Subjects with a history of invasive malignancy within 5 years of study entry.
* History of allergic reactions to α-lactalbumin, human milk (excluding lactose intolerance), zymosan, or other agents used in this study.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Subjects with known hyperprolactinemia
* Subjects being treated with drugs known to cause hyperprolactinemia
* Subjects having lactated within 6 months of study start (first dose of vaccine).

Pembrolizumab Cohort:

* All exclusion criteria for the pembrolizumab cohort will be the same as the TNBC cohort as outlined above, with the exception of: Failure to recover from the toxicity of the previous therapy to CTCAE Grade 0-1, except for:

  * Alopecia
  * Grade 2 neuropathy, or,
  * Grade 2 or 3 decreased lymphocyte count/lymphopenia (only in the pembrolizumab cohort in patients having received radiation therapy within 6 months of study enrollment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Treatment Cohort MTD of α-lactalbumin vaccine | Day 84
  MTD of an α-lactalbumin vaccine in participants with operable triple-negative breast cancer
Preventative Cohort MTD of α-lactalbumin vaccine | Day 84
  MTD of an α-lactalbumin vaccine in participants at risk for TNBC who are scheduled for prophylactic double mastectomy.
Pembrolizumab Cohort of α-lactalbumin vaccine | Day 84
  MTD of an α-lactalbumin vaccine in participants who are receiving adjuvant pembrolizumab following initial TNBC treatment.

SECONDARY OUTCOMES:
Treatment Cohort Lowest Immunologic Dose (LID) of α-lactalbumin vaccine | Day 84
  LID of α-lactalbumin vaccine in participants with operable triple-negative breast cancer, based on ELISPOT assays to assess the ability to induce a pro-inflammatory T cell response consistent with tumor protection. This assessment will be determined using the ELISPOT assay to determine peripheral blood frequencies of T cells that produce interferon-gamma (IFNγ; type-1) and IL-17 (type-17) in response to recombinant human α-lactalbumin
Preventative Cohort Lowest Immunologic Dose (LID) of α-lactalbumin vaccine | Day 84
  LID of α-lactalbumin vaccine in participants at risk for TNBC who are scheduled for prophylactic double mastectomy, based on ELISPOT assays to assess the ability to induce a pro-inflammatory T cell response consistent with tumor protection. This assessment will be determined using the ELISPOT assay to determine peripheral blood frequencies of T cells that produce interferon-gamma (IFNγ; type-1) and IL-17 (type-17) in response to recombinant human α-lactalbumin
Pembrolizuman Cohort Lowest Immunologic Dose (LID) of α-lactalbumin vaccine | Day 84
  LID of α-lactalbumin vaccine in participants who are receiving adjuvant pembrolizumab following initial TNBC treatment, based on ELISPOT assays to assess the ability to induce a pro-inflammatory T cell response consistent with tumor protection. This assessment will be determined using the ELISPOT assay to determine peripheral blood frequencies of T cells that produce interferon-gamma (IFNγ; type-1) and IL-17 (type-17) in response to recombinant human α-lactalbumin

CONTACTS AND LOCATIONS:
Overall Officials: George T Budd, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Yes, the data will be shared with the FDA, the Department of Defense (DOD), and Anixa Biosciences who has negotiated rights to the drug, and any pharmaceutical partner who may wish to negotiate rights to the drug. All below may be shared, with patient data anonymized
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available during the course of the trial and indefinitely thereafter.
Access Criteria: The data will be available to the FDA and DOD. Otherwise, a confidentiality agreement will need to be in place.